CLINICAL TRIAL: NCT02440776
Title: Pathway CH S&E Registry: Data Collection on the ATI Neurostimulation System: SPG Stimulation for Cluster Headache - ATI Neurostimulation System is Branded Internationally as Pulsante™ Microstimulator System
Brief Title: Pathway CH S&E Registry
Acronym: SER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-010
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Monitor the safety and performance of the Pulsante Microstimulator System.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets CE marked labeling for cluster headache.
2. Patient has the ability to read, comprehend and reliably record information as required by the Protocol.
3. Patient is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

1. Patient has other significant pain problem that might confound the study assessments in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who meet the CE marked labeling for cluster headache for the Pulsante Microstimulator System
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-05-13 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of all device/procedure related Adverse Events | Through five years post implant
  Outcome will be assessed at Implant, 3, 6, 9, 12, 18, 24, 36, 48 and 60 months post implant.

SECONDARY OUTCOMES:
Acute response to therapy | Through five years post implant
  Outcome will be assessed at 3, 6, 9, 12, 18, 24, 36, 48 and 60 months post implant.

CONTACTS AND LOCATIONS:
Locations (9):
- Rigshospitalet Neurocenter, Glostrup Municipality, Denmark
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Klinik und Poliklinik für Neurologie, Dresden
  - Heinrich-Heine-University, Düsseldorf
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinik für Schmerztherapie, Rotes Kreuz Krankenhaus, Hansteinstr. 29, Kassel
  - Neurologie + Kopfschmerzzentrum Münchner Freiheit, Munich
- Neurologiska Kliniken-Karolinska UniversitetssjukhusetSolna, Stockholm, Sweden
- University Hospital Zurich, Klinik f. Neurologie, Frauenklinikstr. 26, Zurich, Switzerland
- The Walton Center, Liverpool, United Kingdom